CLINICAL TRIAL: NCT06453109
Title: Towards Treatment of the Complex Patient: Investigations of Low-intensity Focused Ultrasound
Brief Title: Focused Ultrasound for the Complex Patient
Acronym: LIFU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1777666; UG3DA059407 (NIH)
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use Disorder; Chronic Back Pain; Anxiety
Keywords: anxiety disorders; oud; opiate use disorder; opioid; back pain; chronic back pain; opioid use; opioid abuse; opioid disorder; low intensity focused ultrasound; transcranial ultrasound
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders; Back Pain

STUDY DESIGN:
Intervention Model Description: within subject, randomized, double-blind, sham-controlled trial
Who Masked: Participant, Investigator
Masking Description: The Sham condition will be conducted using an interface which does not allow ultrasound energy to pass from the transducer to the target. The administration of LIFU/sham will be conducted in a double-blind fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LIFU/Sham (Other): double-blind, sham-controlled, crossover study in N=25 individuals with opiate use disorder, anxiety, and chronic back pain
  Interventions: Device: low intensity focused ultrasound (LIFU)
- Sham/LIFU (Other): double-blind, sham-controlled, crossover study in N=25 individuals with opiate use disorder, anxiety, and chronic back pain
  Interventions: Device: low intensity focused ultrasound (LIFU)

INTERVENTIONS:
Device: low intensity focused ultrasound (LIFU) — Low-intensity focused ultrasound (LIFU) provides an energy source with millimeter resolution that can be focused anywhere in the brain safely and effectively for non-invasive and transient neuromodulation. LIFU is an important advance and of great significance for brain-mapping efforts, diagnostics, and therapies in neuroscience and particularly promising for addiction therapy as it provides unprecedented non-surgical access to the brain regardless of depth.
  Much lower intensities of focused ultrasound (LIFU) are used so that tissue damage does not occur, but neural activity can be modulated. LIFU utilizes acoustic energy at much lower levels to affect tissue by mechanical effects.

SUMMARY:
The goal of this clinical trial is to to inhibit the anterior insula (AI) with low intensity focused ultrasound (LIFU) to determine the causal role for the AI in pain processing, anxiety, and opiate cue-induced craving. The main question[s] it aims to answer are:

* the safety and tolerability of LIFU delivered bilaterally to AI compared to sham stimulation in individuals with opiate use disorder (OUD), anxiety, and chronic back pain
* the effects of LIFU vs sham on measures of pain processing, anxiety symptoms, and opiate cue-induced craving

Participants will undergo anatomical MRI, neurological assessment, clinical assessment and patient query to assess the safety and tolerability of LIFU vs sham.

DETAILED DESCRIPTION:
Opioid use disorder with co-morbid chronic pain and anxiety is a clinical triad associated with the highest risk of opiate overdose deaths. Co-occurrence of these three disorders amplifies symptoms of each and results in poorer treatment outcomes. There are shared neurobiological substrates for these disorders such as reward processing and stress response. The anterior insula (AI) is a brain region involved in these processes as well as in clinical disorder of pain, addiction, and anxiety. The AI is upregulated in pain, addiction and anxiety disorders and is therefore a potential therapeutic target for neuromodulation. Low-intensity focused ultrasound (LIFU) is a noninvasive method to inhibit cortical and deep brain regions. LIFU can reach deep brain regions such as the AI with spatial specificity, unlike traditional noninvasive neuromodulation methods which lack spatial specificity and depth penetration. LIFU can selectively target the insula and its subregions and provides a potentially transformative method to reduce symptoms of pain, opiate craving, and anxiety in a complex patient population such as co-morbid chronic pain, anxiety, and opioid use disorder. In this study, the investigators will administer one session of inhibitory LIFU to the AI in individuals with opiate use disorder, chronic back pain, and anxiety disorders (generalized anxiety disorder, post-traumatic stress disorder, or social anxiety disorder)]. The aim of this phase of the study is to establish that LIFU vs sham LIFU to AI is safe and well tolerated as measured by adverse events, clinical evaluation and repeated structural brain magnetic resonance imaging scans. The investigators will also gather preliminary data on the effect of LIFU to AI on opiate cue-induced craving and laboratory measures of central sensitization(CS) which occurs with pain chronicity such as temporal summation of pain and conditioned pain modulation. There is a need for improved treatments for complex patients such as co-morbid chronic back pain, anxiety, and opioid use disorder beyond combining treatments for each disorder. LIFU provides an ability to transiently and selectively inhibit AI to determine its causal role in co-morbid chronic back pain, anxiety, and opioid use disorder symptoms which then may lead to improved treatments for this clinical triad which is associated with poor treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-75 years
2. Current diagnosis of Chronic Back Pain as defined by pain duration of at least three months, with back pain being an ongoing problem for at least half the days of the last six months.
3. Have evidence of central sensitization (CS) as measured by the Widespread Pain/Symptom Severity Index (WPSSI) with a score of Widespread Pain Index (WPI) ≥ 7 and Symptom Severity (SS) ≥ 5 or WPI = 3-6 and SS ≥ 9.
4. Participants must rate pain intensity at 4/10 or greater on the Brief Pain Inventory-Short Form (BPI-SF)
5. Meet the DSM-5 criteria for current opiate use disorder as diagnosed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition.
6. Be in treatment for OUD including buprenorphine or methadone.
7. Meet the DSM-5 criteria for a current anxiety disorder: generalized anxiety disorder, post-traumatic stress disorder or social anxiety disorder as diagnosed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition(DSM-5).

Exclusion Criteria:

1. Evidence of neuropathic pain
2. Current DSM-5 substance use disorder other than OUD, tobacco use disorder
3. Current DSM-5 diagnosis of schizophrenia or schizo-affective disorder
4. Pregnant or breastfeeding
5. Daily use of benzodiazepines or opiates (other than buprenorphine or methadone)
6. History of seizures, neurologic disorders, including cerebrovascular disease, history of stroke, brain surgery, brain tumor, multiple sclerosis, or neurodegenerative diseases. They will not have history of metastasizing cancers, inflammatory disorder: rheumatoid arthritis, polymyalgia rheumatica, scleroderma, lupus or polymyositis, unintended weight loss of 20 pounds or more in the last year, or cauda equina syndrome.
7. Ferromagnetic implants or other contraindications for MRI
8. Unstable medical conditions such as congestive heart failure, unstable angina, poorly controlled arrhythmia active systemic infection end stage renal disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | immediately prior to 1 session low-intensity focused ultrasound (LIFU) and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post sham
  number of adverse events

SECONDARY OUTCOMES:
Heart rate variability | immediately prior to 1 session low-intensity focused ultrasound (LIFU) and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post sham
  Continuous heart rate variability monitoring
Pain threshold | immediately prior to 1 session low-intensity focused ultrasound (LIFU) and within 1 hour post LIFU; immediately prior to 1 session sham and with in 1 hour post sham
  Numeric Pain Rating Scale (NPRS) Score: 0-10 0 = 'No pain' 10 = 'Worst pain imaginable'

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Lee, MD, Principal Investigator — Washington D.C. Veterans Affairs Medical Center
Locations (1):
- Washington DC Veterans Affairs Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
behavioral and imaging data
Supporting Information: SAP, Analytic Code
Time Frame: data will be available after analysis of primary and secondary outcomes are completed